CLINICAL TRIAL: NCT05415319
Title: Relation of Emotion Regulatory Behaviors in Early Childhood to Cognitive Emotion Regulation Strategies in Middle Childhood and Pre-Adolescence
Brief Title: Emotion Regulation Strategies in Toddlerhood and Middle Childhood
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded.
Sponsor: Miami University (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KielR032022
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: All children will experience brief standardized laboratory tasks according to the same protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotion regulation observation in middle childhood/pre-adolescence (Other): All participants will engage in brief laboratory tasks that are designed to elicit a brief experience of emotion/uncertainty.
  Interventions: Behavioral: Laboratory tasks in middle childhood/pre-adolescence

INTERVENTIONS:
Behavioral: Laboratory tasks in middle childhood/pre-adolescence — Children will watch a 2-minute clip from a live-action movie and complete Storytelling and Mask tasks from the Laboratory Temperament Assessment Battery.

SUMMARY:
This study will examine the relation between behavioral emotion regulation (ER) strategies at toddler age 3 to cognitive ER strategies in middle childhood/pre-adolescence as part of an ongoing longitudinal study of children's typical development. Aim 1 is to test whether self-soothing/caregiver-focused and distraction behavioral ER strategies at child age 3 predict avoidant and engaging cognitive ER strategies, respectively, at a follow-up assessment to be completed when children are 8-14 years old. In a completed wave of data collection, children's ER behaviors were elicited in laboratory tasks characterized by novelty and uncertainty at age 3. Avoidant and engaged cognitive ER strategies will be assessed by children's self-report, parent-report, and interviews with children after they engage in new laboratory tasks characterized by uncertainty. Hypothesis 1a: Self-soothing/caregiver-focused toddler behavioral ER strategies will predict avoidant cognitive strategies in middle childhood/pre-adolescence. Hypothesis 1b: The toddler behavioral ER strategy of distraction will predict engaged cognitive ER strategies in middle childhood/pre-adolescence. To provide additional developmental information, Aim 2 is to test whether child age at the follow up assessment (ranging 8-14 years) moderates the relation between behavioral ER strategies at age 3 and cognitive emotion regulatory strategies in middle childhood/pre-adolescence. Hypothesis 2: Because older children will have undergone more development underlying cognitive ER strategies, relations specified in Hypotheses 1a and 1b will strengthen across older ages. Finally, the Exploratory Aim is to test theoretically-supported individual (i.e., temperament) and environmental (i.e., family emotional environment) variables as potential mediators or moderators of the relation between behavioral ER strategies at age 3 and cognitive ER strategies in middle childhood-preadolescence. The investigators expect inhibited temperament to be involved in the link between behavioral ER strategies and avoidant cognitive ER strategies, effortful control to be involved in the link between behavioral ER strategies and engaged cognitive ER strategies, and the emotional family environment to be involved in linking behavioral ER strategies to both avoidant and engaged ER strategies.

DETAILED DESCRIPTION:
Children (8 to 14 years) will be invited to come to a 1.5 hour laboratory assessment with a parent (most likely, mothers). We will gather parent-reported and children's self-reported avoidant and engaged cognitive ER strategies, worded with third or first person, respectively. "Short form" versions will be used to reduce burden for children. The Emotion Regulation Questionnaire for Children and Adolescents provides a 6 item reappraisal scale and a 4 item expressive suppression scale. The Avoidance and Fusion Questionnaire for Youth - Short Form provides an 8-item measure of experiential avoidance. The extended version of the Children's Response Styles Questionnaire provides a 5 item scale of problem-solving (also, "reflection") and a 5 item scale of rumination (also, "brooding"). Mothers will complete the Children's Responses to Feelings Checklist, which asks about these ER strategies in response to specific emotions, to examine specificity to uncertainty/fear.

The investigators will also assess "in-vivo" use of cognitive ER strategies by using an ER strategy interview after children experience uncertainty via laboratory procedures. Children will watch a 2-minute clip from a live-action movie validated to elicit emotion in the domain of uncertainty with school-aged children. The primary experimenter will interview the child about the cognitive ER strategies they used using open-ended questions with subsequent prompts to allow reports of multiple strategies. The primary experimenter will then ask closed-ended (yes/no) interview questions about each of the cognitive ER strategies of focus. Children will also complete two 5 minute tasks from the Laboratory Temperament Assessment Battery - Middle Childhood Version with established reliability and validity in the domain of uncertainty. In the "Storytelling" task, the experimenter will instruct the child to stand and tell a story about the previous day in front of them and an unfamiliar research assistant (RA), enacting a series of standardized pauses and prompts until the child indicates they are finished. In the "Mask" episode, the child enters a room to see an adult RA wearing a mask resembling a disfigured face. The RA completes a standardized script of statements and pauses, finally taking off the mask and engaging the child in a friendly manner. The primary experimenter will repeat the ER strategy interview for the tasks. Auxiliary ER-relevant outcomes may supplement the primary focus on cognitive ER strategies. Behavioral tasks (Storytelling, Mask) can be coded for behavioral ER strategies (distraction, self-soothing, bids to experimenter). The investigators possess the necessary equipment and software for recording and analysis of children's ECG and respiration to serve as physiological indicators of ER. As an additional indicator of family emotional environment, the child and mother will be prompted to converse about the activities in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Family participated in previous phases of this ongoing longitudinal study
* Child was 35-42 months old for the age 3 assessment (pre-existing data)
* Child is between 8 and 14 years of age for proposed data collection
* Mothers were older than 18 years of age at original enrollment (pre-existing data).
* Mothers were able to complete study procedures in English.

Exclusion Criteria:

* Informed consent/assent is declined
* Child diagnosed with a developmental disability or chronic health condition related to deviations in expected emotional development.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire for Children and Adolescents | 3 minutes (at 1.5 hour laboratory visit)
  Parent- and child self-report versions of this survey measure, including 6-item Reappraisal subscale and 4-item Expressive Suppression subscale
Avoidance and Fusion Questionnaire for Youth-Short Form | 2 minutes (at 1.5 hour laboratory visit)
  Parent- and child self-report versions of this survey measure, which provides an 8-item subscale of Experiential Avoidance
Children's Response Styles Questionnaire | 2 minutes (at 1.5 hour laboratory visit)
  Parent- and child self-report versions of this survey measure, which provides a 5-item subscale of Problem-Solving/Reflection, and a 5-item subscale of Rumination/Brooding.

SECONDARY OUTCOMES:
Electrocardiogram | 1.5 hours over the course of laboratory visit
  Respiratory sinus arrhythmia (RSA) will be derived as a metric of variance in interbeat intervals at rate of respiration, exhibited during laboratory tasks
Children's Responses to Feelings Checklist | 2 minutes (at 1.5 hour laboratory visit)
  Present versus absent responses will indicate parents' perception that children use particular emotion regulatory strategies within specific emotional domains (happiness, anger, fear/uncertainty)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Kiel Luebbe, Ph.D., Principal Investigator — Miami University
Locations (1):
- Miami University Department of Psychology, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified and processed data will be posted to Open Science Framework. No identifying information will be shared. Final version of data (e.g., behavioral coding composites, survey scores) reported in manuscripts will be shared.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be posted towards the end of the grant period (months 21-24), should funding be received. Data will be available indefinitely.
Access Criteria: Academic affiliation